CLINICAL TRIAL: NCT05732701
Title: Algorithm-based Tailoring of Dual Antiplatelet Therapy to Improve Outcomes Following Percutaneous Coronary Interventions
Acronym: TAILOR-DAPT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TAILOR-DAPT
Record Dates: First submitted 2023-02-08; First posted 2023-02-17 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Percutaneous Coronary Intervention; Platelet Aggregation Inhibitors; Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Single-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Algorithm-guided DAPT duration
  Interventions: Other: Algorithm-guided DAPT duration
- Standard (Active Comparator): Standard-of-care DAPT duration
  Interventions: Other: Standard-of-care DAPT duration

INTERVENTIONS:
Other: Algorithm-guided DAPT duration — PRECISE-DAPT score ≥25
  * Chronic Coronary Syndromes (CCS): Aspirin + clopidogrel for 1 month, followed by clopidogrel monotherapy
  * Acute Coronary Syndromes (ACS): Aspirin + ticagrelor for 1 month, followed by ticagrelor monotherapy
  PRECISE-DAPT score <25:
  * Non-complex CCS: Aspirin + clopidogrel for 6 months, followed by clopidogrel monotherapy
  * Non-complex ACS: Aspirin + potent P2Y12 inhibitor for 6 months, followed by potent P2Y12 inhibitor monotherapy
  * Complex CCS or ACS: Aspirin + P2Y12 inhibitor for 12 months, followed by P2Y12 inhibitor monotherapy (potent P2Y12 inhibitor mandatory for ACS)
  Arms: Intervention
Other: Standard-of-care DAPT duration — DAPT strategy at the operators´ discretion in accordance with applicable guidelines
  Arms: Standard

SUMMARY:
The use of aspirin combined with a P2Y12 inhibitor (dual antiplatelet therapy, DAPT) represents the standard of care for patients undergoing percutaneous coronary intervention (PCI) with stent implantation. The TAILOR-DAPT trial aims to investigate the benefits of a score-based decision-making algorithm to guide DAPT duration compared to a standard-of-care DAPT duration without the use of risk scores in patients undergoing PCI.

DETAILED DESCRIPTION:
Background:

The use of aspirin combined with a P2Y12 inhibitor (dual antiplatelet therapy, DAPT) represents the standard of care for patients undergoing percutaneous coronary intervention (PCI) with stent implantation. European guidelines recommend to implement risk scores to guide the duration of DAPT after stent implantation (class IIb, level of evidence A). However, its adoption rate remains exceedingly low in daily clinical practice in part due to the lack of direct evidence obtained from a randomized controlled trial supporting this strategy.

Aim:

Using a pragmatic study-design, the investigators aim to determine the efficacy and safety of an algorithm-guided strategy for DAPT duration compared to a standard-of-care DAPT without the use of risk scores in patients undergoing PCI with stent implantation.

Methodology:

This investigator-initiated, single-blind, randomized trial will include a total of 2788 patients aged ≥18 years undergoing PCI with stent implantation. Main exclusion criteria are peri-procedural complications potentially affecting DAPT duration. The study will be nested into a well-running registry to minimize study-related costs (pragmatic trial approach). Patients will be randomized to an algorithm-guided DAPT group or a standard-of-care DAPT group in a 1:1 fashion. In the algorithm-guided group, DAPT duration will be determined according to the PRECISE-DAPT score (≥25 or <25), PCI complexity, and clinical presentation (acute or chronic coronary syndromes). In the standard-of-care DAPT group, treatment duration is at the operator's discretion. The primary endpoint is a composite of net adverse clinical events (NACE) defined as all-cause death, spontaneous myocardial infarction, stroke, definite stent thrombosis or Bleeding Academic Research Consortium (BARC) 2, 3, or 5 bleeding at 1 year.

Potential significance:

This will be the first study evaluating the impact of a score-based decision-making algorithm integrating bleeding and ischemic risks for DAPT duration among patients undergoing PCI. The hypothesis is that the proposed simple decision-making algorithm minimizes bleeding risk and maximizes ischemic benefit compared to a standard-of-care DAPT regimen. Prospective data obtained from a pragmatic randomized controlled trial embedded into an on-going, well-managed PCI registry database may further enhance the adoption rate of such a strategy in clinical practice.

ELIGIBILITY:
Inclusion Criteria:

1. PCI with drug eluting stent (DES) implantation
2. Age ≥18 years
3. Ability to sign informed consent before any study-specific procedure

Exclusion Criteria:

1. Planned staged PCI (Patients can be enrolled after complete coronary revascularization with no remaining lesions intended for treatment. Patients who have or develop an indication for percutaneous valve intervention can undergo treatment 30 days after full coronary revascularization)
2. Indication for oral anticoagulation
3. Peri-procedural complication which affects DAPT regimen based on the operator's opinion (e.g. untreated flow-limiting angiographic complication, intraprocedural stent thrombosis, persistent vessel occlusion/no-reflow at the end of the procedure, major side-branch occlusion, puncture-site related or other relevant bleeding)
4. Treatment for stent thrombosis at qualifying PCI or within 1 year prior to qualifying PCI
5. Active bleeding requiring medical attention at qualifying PCI
6. The presence of hemodynamic instability (persistent systolic blood pressure below 90mmHg, continuous infusions of catecholamines, clinical signs of hypoperfusion and/or use of percutaneous left ventricular assist devices)
7. Life expectancy less than 1 year
8. Women of childbearing potential (i.e. fertile, following menarche and until becoming post-menopausal unless permanently sterile)
9. Planned surgery within the next 3 months
10. Contraindication or known allergy against aspirin or P2Y12 inhibitors (clopidogrel, ticagrelor, and prasugrel)
11. Participation in a drug trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2788 (Estimated)
Dates: Start 2023-06-27 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Net adverse clinical events (NACE) | 1 year
  All-cause death, spontaneous myocardial infarction, definite stent thrombosis, stroke or Bleeding Academic Research Consortium (BARC) 2, 3 or 5 bleeding

SECONDARY OUTCOMES:
Major adverse cardiovascular events (MACE) | 1 year
  Cardiovascular death, spontaneous myocardial infarction, definite stent thrombosis or stroke
Major or clinically relevant non-major bleeding | 1 year
  Bleeding Academic Research Consortium (BARC) 2, 3 or 5 bleeding
Major bleeding | 1 year
  Bleeding Academic Research Consortium (BARC) 3 or 5 bleeding
Any Bleeding Academic Research Consortium (BARC) bleeding | 1 year
All-cause death | 1 year
Cardiovascular death | 1 year
Myocardial infarction | 1 year
Spontaneous myocardial infarction | 1 year
Target lesion failure | 1 year
  Cardiac death, target-vessel myocardial infarction or target lesion revascularization
Target vessel revascularization | 1 year
Target vessel myocardial infarction | 1 year
Target lesion revascularization | 1 year
Non-target vessel revascularization | 1 year
Any revascularization | 1 year
Definite stent thrombosis | 1 year
Stroke | 1 year
Transient ischemic attack | 1 year
Adherence to DAPT | 1 year
  According to the TAILOR-DAPT modified Non-adherence Academic Research Consortium (NARC) classification
Adherence to DAPT | 1 year
  According to the traditional classification (Adherent≥80% of the time from randomization to intended DAPT cessation date)

OTHER OUTCOMES:
Net adverse clinical events (NACE) | 24 months
  All-cause death, spontaneous myocardial infarction, definite stent thrombosis, stroke or Bleeding Academic Research Consortium (BARC) 2, 3 or 5 bleeding

CONTACTS AND LOCATIONS:
Overall Officials: Lorenz Räber, MD, PhD, Study Chair — Department of Cardiology, Bern University Hospital, Bern, Switzerland; Miklos Rohla, MD, PhD, Principal Investigator — Department of Cardiology, Bern University Hospital, Bern, Switzerland
Locations (3):
- University Clinical Center of the Republic of Srpska, Banja Luka, Bosnia and Herzegovina
- UOC Cardiologia San Giovanni Addolorata Hospital, Roma, Italy
- Department of Cardiology, Bern University Hospital, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No